CLINICAL TRIAL: NCT00003934
Title: Phase III Randomized Study of Concurrent Tretinoin and Chemotherapy With or Without Arsenic Trioxide (AS2O3) (NSC # 706363) as Initial Consolidation Therapy Followed by Maintenance Therapy With Intermittent Tretinoin Versus Intermittent Tretinoin Plus Mercaptopurine and Methotrexate for Patients With Untreated Acute Promyelocytic Leukemia
Brief Title: Tretinoin, Cytarabine, and Daunorubicin Hydrochloride With or Without Arsenic Trioxide Followed by Tretinoin With or Without Mercaptopurine and Methotrexate in Treating Patients With Acute Promyelocytic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02811; C9710; CDR0000067126; CALGB-C9710; U10CA031946 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Promyelocytic Leukemia (M3); Childhood Acute Promyelocytic Leukemia (M3); Untreated Adult Acute Myeloid Leukemia; Untreated Childhood Acute Myeloid Leukemia and Other Myeloid Malignancies
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute | interventions — Tretinoin; Daunorubicin; Cytarabine; Mercaptopurine; Methotrexate; merphos; Arsenic Trioxide

ARMS (2):
- Arm I (Experimental): Induction: All patients receive oral tretinoin every 12 hours beginning on day 1 until complete response or for a maximum of 90 days. Patients also receive daunorubicin IV on days 3-6 and cytarabine IV continuously on days 3-9.
  Consolidation: All patients achieving CR or PR after completion of tretinoin, proceed to consolidation within 2 weeks of achieving CR or PR, but not prior to 30 days from the start of induction. Patients are randomized to 1 of 2 treatment arms.
  Patients receive oral tretinoin every 12 hours on days 1-7 and daunorubicin IV on days 1-2 or days 1-3, depending on age. Patients may receive an additional course. Treatment begins no earlier than 2 weeks and no later than 4 weeks after hematopoietic recovery.
  Interventions: Drug: tretinoin; Drug: daunorubicin hydrochloride; Drug: cytarabine; Drug: arsenic trioxide
- Arm II (Experimental): Induction: All patients receive oral tretinoin every 12 hours beginning on day 1 until complete response or for a maximum of 90 days. Patients also receive daunorubicin IV on days 3-6 and cytarabine IV continuously on days 3-9.
  Consolidation: All patients achieving CR or PR after completion of tretinoin, proceed to consolidation within 2 weeks of achieving CR or PR, but not prior to 30 days from the start of induction. Patients are randomized to 1 of 2 treatment arms.
  Patients receive oral tretinoin as in arm I above. Patients also receive oral mercaptopurine once a day and oral methotrexate once weekly for up to 1 year.
  Interventions: Drug: tretinoin; Drug: daunorubicin hydrochloride; Drug: cytarabine; Drug: mercaptopurine; Drug: methotrexate; Drug: arsenic trioxide

INTERVENTIONS:
Drug: tretinoin — Given orally
  Other Names: ATRA; Retin-A; TRA
Drug: daunorubicin hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; daunomycin hydrochloride; daunorubicin; RP-13057
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Drug: mercaptopurine — Given IV
  Other Names: 6-mercaptopurine; 6-MP; Leukerin; MP
  Arms: Arm II
Drug: methotrexate — Given IV
  Other Names: amethopterin; Folex; methylaminopterin; Mexate; MTX
  Arms: Arm II
Drug: arsenic trioxide — Given IV
  Other Names: Arsenic (III) Oxide; Arsenic Sesquioxide; Arsenous Acid Anhydride; AS2O3; Trisenox

SUMMARY:
This randomized phase III trial is studying tretinoin and combination chemotherapy to see how well they work compared to tretinoin, combination chemotherapy, and arsenic trioxide in treating patients with acute promyelocytic leukemia that has not been treated previously. Drugs used in chemotherapy, such as daunorubicin, cytarabine, mercaptopurine, methotrexate, and arsenic trioxide, work in different ways to stop cancer cells from dividing so they stop growing or die. Tretinoin may help leukemia cells develop into normal white blood cells. It is not yet known which regimen is more effective for acute promyelocytic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

i. To compare the efficacy (event-free survival) and toxicities of two induction/consolidation therapies for patients with untreated APL: ATRA/ara-C/daunorubicin with or without arsenic trioxide (As2O3).

II. To evaluate the efficacy (disease-free survival) and toxicities of maintenance therapy with intermittent ATRA vs intermittent ATRA plus 6-MP/MTX for patients with APL who achieve a complete response.

III. To explore the relationship between CD56 expression at diagnosis and clinical outcomes.

IV. To evaluate the cardiac toxicity of intensive daunorubicin therapy, as given in this study, to pediatric patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to age (under 15 vs 15 to 60 vs over 60) for the induction phase. Patients are stratified according to age, as in the induction phase, and the consolidation arm (with vs without arsenic trioxide) for the consolidation phase. Patients under age 5 do not receive arsenic trioxide.

Induction: All patients receive oral tretinoin every 12 hours beginning on day 1 until complete response or for a maximum of 90 days. Patients also receive daunorubicin IV on days 3-6 and cytarabine IV continuously on days 3-9.

Consolidation: All patients achieving complete response (CR), or partial response (PR) after completion of tretinoin, proceed to consolidation within 2 weeks of achieving CR or PR, but not prior to 30 days from the start of induction. Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive oral tretinoin every 12 hours on days 1-7 and daunorubicin IV on days 1-2 or days 1-3, depending on age. Patients may receive an additional course. Treatment begins no earlier than 2 weeks and no later than 4 weeks after hematopoietic recovery.

Arm II: Patients receive arsenic trioxide IV over 2 hours daily 5 days a week for 5 weeks. After a 2-week rest, patients receive a second course of arsenic trioxide. Patients then receive tretinoin and daunorubicin as in arm I.

Maintenance: Patients maintaining CR or PR after consolidation therapy proceed to maintenance therapy, beginning no earlier than 2 weeks and no later than 4 weeks after hematopoietic recovery. Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive oral tretinoin every 12 hours for 7 days every other week for 1 year.

Arm II: Patients receive oral tretinoin as in arm I above. Patients also receive oral mercaptopurine once a day and oral methotrexate once weekly for up to 1 year.

Maintenance therapy continues for up to 1 year in the absence of unacceptable toxicity.

Patients are followed every 2 months for 2 years, every 3 months for 1 year, every 6 months for 2 years, and then annually for 5 years.

PROJECTED ACCRUAL: A total of 522 patients (456 adults and 66 pediatric) will be accrued for this study within 4.75 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a clinical diagnosis of acute promyelocytic leukemia (APL) with proof of APL morphology (FAB-M3) confirmed by RT-PCR assay; a patient may be entered prior to completion of RT-PCR studies, but a patient who is subsequently found to be PML-RARα negative and RARα-PML negative will be removed from protocol treatment
* FAB clasification: the aspirate smear must show M3 characteristics and at least 30% of cells must be abnormal promyelocytes with heavy granulation; the overall marrow cellularity must be normocellular or hypercellular; patients with the microgranular variant (M3V) are eligible, and the diagnosis will be based on characteristic morphologic findings (e.g., reniform or bilobed nuclei)
* RT-PCR assay: submission of samples for RT-PCR assays for PML-RARα/RARα-PML transcripts is mandatory; the results do not have to be known prior to initiation of therapy; if the assay is subsequently found to be negative, the patient will be removed from protocol treatment and treated at the discretion of the responsible physician
* Prior treatment: the patient must not have received any systemic definitive treatment for APL, including cytotoxic chemotherapy or retinoids; prior therapy with corticosteroids, hydroxyurea or leukapheresis will not exclude the patient
* Non-pregnant, non-nursing: treatment under this protocol would expose an unborn child to significant risks; patients should not be pregnant or plan to become pregnant while on treatment; women and men of reproductive potential should agree to use an effective means of birth control; there is an extremely high risk of fetal malformation if pregnancy occurs while on ATRA in any amount even for short periods

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 1999-06; Primary Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Response rates | Up to 10 years
Distributions of event-free survival | Up to 10 years
Disease-free survival | Time from the date of the maintenance randomization to relapse or death, assessed up to 10 years
Survival | Up to 10 years
Toxicities for the various therapies graded according to the National Cancer Institute Common Toxicity Criteria (NCI CTC) v2.0 | Up to 30 days after last dose of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bayard Powell, Principal Investigator — Cancer and Leukemia Group B
Locations (2):
- United States (2):
  - Cancer and Leukemia Group B, Chicago, Illinois
  - Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina

REFERENCES:
- [Derived] Powell BL, Moser B, Stock W, Gallagher RE, Willman CL, Stone RM, Rowe JM, Coutre S, Feusner JH, Gregory J, Couban S, Appelbaum FR, Tallman MS, Larson RA. Arsenic trioxide improves event-free and overall survival for adults with acute promyelocytic leukemia: North American Leukemia Intergroup Study C9710. Blood. 2010 Nov 11;116(19):3751-7. doi: 10.1182/blood-2010-02-269621. Epub 2010 Aug 12. PMID 20705755